CLINICAL TRIAL: NCT04795921
Title: Investigating the Sleeping Habits of Patients With Haemophilia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: University of Wuppertal (Other)
Responsible Party: Principal Investigator, PD Dr. Andreas Strauß, specialist for orthopaedics and trauma surgery, University Hospital, Bonn
Other Study IDs: HaemSleep20210208
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-06

CONDITIONS: Sleep Disorder; Psychological; Activity, Motor
MeSH Terms: conditions — Sleep Wake Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with haemophilia: This investigation includes patients with haemophilia of all seventies (mild, moderate, severe), as well as female carriers and patients with Von-Willebrand-Disease (Typ III)
- Healthy controls: The control group consists of adult healthy female and male subjects.

SUMMARY:
This investigation aims to explore sleeping habits in patients with haemophilia.

These patients often suffer from joint pain, which leads to restricted physical activity. Further, many of the patients suffer from psychological strains, such as depression. Both depression and restricted physical activity can result in sleeping disorders. Thus it is aimed to find out which factors and comorbidities do play a role within sleeping habits in patients with haemophilia.

ELIGIBILITY:
Inclusion Criteria:

* adult (≥ 18 years) patients with haemophilia (all severities) or Von-Willebrand-Disease (Typ III)
* female carriers
* signed informed consent

Exclusion Criteria:

* patients with other bleeding disorders
* patients with acute injuries, psychological disorders or Prior surgeries (in the last 6 weeks)
* no signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to include 104 patients with haemophilia as well as 104 age-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Sleeping habits | 15 Minutes
  Questionnaire on sleeping habits (SF/BR B)

SECONDARY OUTCOMES:
Physical activity | 10 Minutes
  Questionnaire on physical activity level (self-developed Questionnaire)
Psychological distress | 10 Minutes
  Health survey of psychological distress (PHQ9)
Kinesiophobia | 5 Minutes
  Tampa Scale of Kinesiophobia (scale 1-5)
Subjective pain perception | 5 Minutes
  Questionnaire on Pain Sensitivity
Adherence to prophylactic treatment | 5 Minutes
  Questionnaire on adherence to prophylactic Treatment (VERITAS-Pro)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Bonn, Bonn, Northrhine Westfalia, Germany

IPD SHARING:
Plan to Share IPD: No
The publication of anonymous patient data is not allowed by informed consent.